CLINICAL TRIAL: NCT03119012
Title: SMart Angioplasty Research Team: Comparison Between P2Y12 Inhibitor MonotHerapy and Dual Antiplatelet Therapy in Patients UndergOing Implantation of Coronary BiorEsorbable Scaffold II: (SMART-CHOICE II) Trial
Brief Title: P2Y12 Inhibitor Monotherapy Versus Extended DAPT in Patients Treated With Bioresorbable Scaffold
Acronym: SMART-CHOICEII
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: cannot use bioabsorbable scaffold
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHOICEII16453143
Record Dates: First submitted 2017-04-01; First posted 2017-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Stents; Atherosclerosis
Keywords: Bioresorbable scaffold; Dual antiplatelet therapy; P2Y12 receptor inhibitor; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Clopidogrel; Ticagrelor; Aspirin

STUDY DESIGN:
Intervention Model Description: Prospective, open label, two-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P2Y12 receptor inhibitor monotherapy arm (Active Comparator): In patients who do not occur a MACCE until 12-month after BRS implantation, P2Y12 receptor inhibitor monotherapy arm will be received clopidogrel 75mg qd or ticagrelor 60mg bid during follow-up period (24 months after randomization).
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor
- Extended DAPT arm (Active Comparator): In patients who do not occur a MACCE until 12-month after BRS implantation, Extended DAPT arm will be received aspirin 100mg qd plus P2Y12 receptor inhibitor (clopidogrel 75mg qd or ticagrelor 60mg bid) during follow-up period (24 months after randomization).
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — 75mg/day
  Other Names: Clopidogrel or its generic
Drug: Ticagrelor — 120mg/day
  Other Names: Brillinta
Drug: Aspirin — 100mg/day
  Other Names: Any commercially available aspirin
  Arms: Extended DAPT arm

SUMMARY:
This study aimed to compare the efficacy and safety of P2Y12 inhibitor monotherapy versus extended dual antiplatelet therapy (DAPT) following 12-month of DAPT in patients undergoing percutaneous coronary intervention (PCI) with bioresorbable scaffold (BRS)

DETAILED DESCRIPTION:
After the development of second generation drug-eluting stent (DES), clinical outcomes including in-stent restenosis have been dramatically improved in patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) compared with bare metal stent or first generation DES era. However, interventional cardiologist still concern about late adverse cardiac events including stent thrombosis (ST) in patients who received implantation of permanent metallic stent. Bioresorbable scaffold (BRS) have been developed to provide mechanical support and drug-delivery function similar to those of DES for approximately 1 year, followed by complete bioresorption over several years. It has the advantages of reducing the risk of late ST and maintaining of normal vascular function because these novel devices are expected to leave no permanent materials within the vessel. Although there was no significant difference from previous randomized controlled studies for evaluating the clinical outcomes at 1-year between BRS and DES, recently documented ARSORB II trial, which compared 3-year outcomes between BRS and DES, show that patients treated with BRS had a higher risk of device-oriented composite endpoint mainly driven by target vessel myocardial infarction (MI) compared to those with DES. In addition, in several case reports, the late ST after discontinuation of dual anti-platelet therapy (DAPT) was reported in patients who underwent BRS implantation. Therefore, the efficacy of extended DAPT and needs for optimal DAPT duration in patients treated with BRS have been emerged. In the DAPT study, randomized controlled trial including approximately 10,000 patients, DAPT beyond 1 year after placement of a DES, as compared with aspirin therapy alone, significantly reduced the risks of major adverse cardiovascular and cerebrovascular events (MACCE) and ST. However, extend use of DAPT increases bleeding risk and cost. Endoscopic, dental, and surgical procedures are often delayed due to extended DAPT, which may affect the patient's quality of life. In addition, there was no significant difference in all-cause mortality between extended DAPT and aspirin monotherapy in the DAPT study because of increased bleeding risk in extended DAPT group. Therefore, to determine the optimal or minimal necessary duration of DAPT is very important. The other important issue is that which antiplatelet agent is more appropriate after DAPT. In CAPRIE (Clopidogrel versus Aspirin in Patients at Risk of Ischaemic Events) trial, clopidogrel showed a superior efficacy in preventing ischemic events compared with aspirin and the incidence of gastrointestinal bleeding was significantly lower with clopidogrel than with aspirin. Moreover, clopidogrel monotherapy was associated with a reduced risk of ischemic events without increased bleeding risk compared with aspirin monotherapy in patients receiving DES after 12-month DAPT. However, current guidelines still recommend aspirin monotherapy after 6-12 months of DAPT in patients treated with DES, there were no data for evaluating the optimal duration of DAPT and preferred choice of monotherapy in patients treated with BRS. Through results of previous studies, the authors postulated that P2Y12 antagonist monotherapy, which might have superior ability to prevent ischemic event compared to aspirin monotherapy, had similar risk of ischemic events with lower risk of bleeding complication compared with extended DAPT in patients who received BRS implantation with 12-month DAPT. Therefore, in the SMART-CHOICE II trial, we will test noninferiority of P2Y12 antagonist monotherapy compared with aspirin plus P2Y12 antagonist after 12-month of DAPT in patients treated with BRS.

Stratification: presence of diabetes mellitus, clinical presentation (acute coronary syndrome), type of P2Y12 inhibitor (clopidogrel or ticagrelor), and investigational center.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age.
* Patients who do not occur a major adverse cardiac and cerebral events (MACCE) at 12-month after BRS implantation
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving P2Y12 antagonist monotherapy or aspirin plus P2Y12 antagonist and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

* Active bleeding
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
* Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
A composite of death, myocardial infarction, and cerebrovascular events | 36 months after the index procedure
  defined as MACCE

SECONDARY OUTCOMES:
All-cause death | 36 months after the index procedure
  Any death
Cardiac death | 36 months after the index procedure
  ARC definition
Myocardial infarction | 36 months after the index procedure
  ARC definition
Cerebrovascular accident | 36 months after the index procedure
  ischemic and hemorrhagic
target lesion revascularization (TLR) | 36 months after the index procedure
  ischemic driven or all
Target vessel revascularization (TVR) | 36 months after the index procedure
  ischemic driven or all
Any revascularization | 36 months after the index procedure
  ischemic driven or all
Stent thrombosis (ST) | 36 months after the index procedure
  definite or probable ST by Academic Research Consortium (ARC) definition
Bleeding Academic Research Consortium (BARC) bleeding 2,3, or 5 | 36 months after the index procedure
  Safety Endpoints, defined as actionable, overt, and fatal bleeding by BARC definition

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked